CLINICAL TRIAL: NCT06789679
Title: Randomized Phase II Clinical Study of Albumin-Bound Paclitaxel and Gemcitabine With or Without S-1 as First-Line Treatment for Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: Albumin-Bound Paclitaxel and Gemcitabine With or Without S-1 as First-Line Treatment for Advanced Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, LIN YANG, Prof, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC5036
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreatic adenocarcinoma; Advanced; First-Line; Efficacy; Safety
MeSH Terms: interventions — Gemcitabine; Albumin-Bound Paclitaxel; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AG Group (Active Comparator): Albumin-bound paclitaxel：125mg/m2，ivgtt，D1，D8，q3w Gem：1000mg/m2，ivgtt，D1，D8，q3w
  Interventions: Drug: Gemcitabine, albumin-bound paclitaxel
- GAS Group (Experimental): Albumin-bound paclitaxel：125mg/m2，ivgtt，D1，q2w Gem：1000mg/m2，ivgtt，D1，q2w S-1：40-60mg Bid，PO，D1-7，q2w
  Interventions: Drug: Gemcitabine, albumin-bound paclitaxel, S-1

INTERVENTIONS:
Drug: Gemcitabine, albumin-bound paclitaxel, S-1 — Albumin-bound paclitaxel：125mg/m2，ivgtt，D1，q2w Gem：1000mg/m2，ivgtt，D1，q2w S-1：40-60mg Bid，PO，d1-7，q2w
  Arms: GAS Group
Drug: Gemcitabine, albumin-bound paclitaxel — Albumin-bound paclitaxel：125mg/m2，ivgtt，D1，D8，q3w Gem：1000mg/m2，ivgtt，D1，D8，q3w
  Arms: AG Group

SUMMARY:
This study is a prospective, open-label, randomized controlled trial that enrolled previously untreated patients with locally advanced or metastatic pancreatic cancer. Participants were randomly assigned to receive either albumin-bound paclitaxel and gemcitabine, or albumin-bound paclitaxel, gemcitabine, and S-1 as first-line treatment. After patients who met the inclusion criteria signed an informed consent form, the study observed patients from the start of treatment until death, withdrawal of consent, loss to follow-up, or the end of the study. Eligible participants were randomly assigned in a 1:1 ratio to either the albumin-bound paclitaxel and gemcitabine treatment group (AG ) or the albumin-bound paclitaxel, gemcitabine, and S-1 treatment group (GAS). A total of 128 patients were planned for inclusion in the study, with 64 in each treatment group. Baseline data related to demographics, disease, treatment, adverse events, and tumor status were collected by the treating physician during the first visit and follow-up visits. Follow-up visits were conducted according to a fixed schedule, with survival assessed every three months through phone calls, WeChat, or by contacting other physicians. The final visit recorded patient death, withdrawal of consent, loss to follow-up, or the conclusion of the study.

ELIGIBILITY:
Inclusion Criteria:

The participant must voluntarily agree to participate in the study and sign the informed consent form.

The participant must be ≥18 years old on the day of signing the informed consent form.

The participant must have a pathological diagnosis of pancreatic ductal adenocarcinoma (including adenosquamous carcinoma).

The participant must not have received any prior systemic treatment for unresectable locally advanced or metastatic pancreatic cancer.

Note: Patients who have received neoadjuvant/adjuvant/radical chemoradiotherapy or neoadjuvant/adjuvant chemotherapy are eligible only if the time from the end of treatment to the first diagnosis of disease progression/recurrence is at least 6 months.

The participant must have measurable lesions according to RECIST 1.1 criteria. If there is only one measurable lesion at baseline, it must not have been previously irradiated or there must be evidence of significant progression since the end of radiotherapy.

The participant must have an ECOG performance status score of 0-2. The participant must have a life expectancy of more than 3 months. The participant must be able to take oral chemotherapy. The participant must meet the required organ function criteria before inclusion.

Female participants of childbearing potential or male participants with partners of childbearing potential must agree to use highly effective contraception starting 7 days before randomization and continue until 24 weeks after treatment initiation. Female participants must have a negative serum pregnancy test within 7 days prior to randomization.

Exclusion Criteria:

Participants with untreated active brain metastases or leptomeningeal metastasis. If brain metastasis has been treated and the disease is stable (with stable imaging for at least 4 weeks prior to randomization and no new neurological symptoms), they may be included.

Participants with untreated spinal compression fractures. Treated spinal compression fractures must be stable for at least 2 weeks before randomization.

Participants who have previously received systemic treatment for unresectable locally advanced or metastatic pancreatic cancer.

Note: Participants who have received neoadjuvant/adjuvant/radical chemoradiotherapy or neoadjuvant/adjuvant chemotherapy are excluded if the time from the end of treatment to disease progression/recurrence is less than 6 months.

Participants with high risk of gastrointestinal or abdominal bleeding. Participants with uncontrolled cancer pain (e.g., requiring escalation of analgesics) at the time of enrollment.

Participants who have received chemotherapy, small molecule inhibitors, immunotherapy (such as interleukins, interferons, or thymosin), or other anti-cancer treatments within 28 days before enrollment, or who have used traditional Chinese medicine with anti-cancer indications within 14 days before enrollment.

Participants who have had major surgery within 28 days before enrollment (excluding diagnostic biopsies such as EUS-FNB or percutaneous liver biopsy).

Participants who have received radical radiation therapy within the last 3 months. Palliative radiation therapy is allowed if administered at least 2 weeks prior to the start of the study treatment.

Participants with a history of another malignancy within the last 5 years, except for treated basal cell carcinoma, squamous cell carcinoma of the skin, non-invasive bladder cancer, or cured prostate/cervical/breast cancer.

Participants with uncontrolled comorbidities, including but not limited to:

Active HBV or HCV infection. Note: Participants with positive HBsAg and/or HCV antibodies must undergo HBV-DNA and/or HCV-RNA testing. Eligible participants must have HBV-DNA ≤500 IU/mL (or ≤2000 copies/mL) and/or HCV-RNA negative.

Known HIV infection or AIDS history. Active syphilis. Active tuberculosis. Active infections. Uncontrolled hypertension, symptomatic heart failure (NYHA II-IV), unstable angina, myocardial infarction within the last 6 months, or QTc prolongation or arrhythmia risk.

Note: Participants with baseline QTc >470 msec (female) / 450 msec (male), hypokalemia, long QT syndrome, resting heart rate >100 bpm in atrial fibrillation, or severe valvular heart disease are excluded.

Active bleeding. Participants whose toxicity from prior anti-cancer treatments has not recovered to CTCAE ≤1 (except for alopecia, which is allowed at any grade, and peripheral neuropathy, which must have recovered to ≤2).

Breastfeeding women. Other conditions that, in the opinion of the investigator, may affect the participant's safety, compliance, or the reliability of the study results, including but not limited to psychiatric disorders, moderate to severe ascites, pleural effusion, pericardial effusion, etc.

Vulnerable populations, including but not limited to those with cognitive impairments, critically ill patients, minors, pregnant women, students/subordinates of the investigator, employees of the study institution or sponsor, and other individuals who may not be able to provide informed consent or comply with the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 1 year

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 1 year
Overall Survival (OS) | 2 years
Progression-free survival(PFS) | 1 year
Disease Control Rate(DCR) | 1 year
Duration of Response (DOR) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lin Yang, Prof, Principal Investigator — LIN YA Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Chaoyang District, China

IPD SHARING:
Plan to Share IPD: No